CLINICAL TRIAL: NCT01368900
Title: Evaluation of the Ulthera® System for Obtaining a Reduction of Wrinkles Around the Eyes
Brief Title: Reducing Wrinkles Around the Eyes Using the Ulthera® System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-111
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2013-09

CONDITIONS: Periorbital Wrinkles
Keywords: Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ulthera System Treatment (Experimental): Ulthera treatment to the upper face.
  Interventions: Device: Ulthera® System treatment

INTERVENTIONS:
Device: Ulthera® System treatment — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy

SUMMARY:
The purpose of this prospective, multi-center, single treatment study is to evaluate the clinical outcomes associated with the non-invasive treatment to reduce wrinkles around the eyes utilizing the Ulthera® System to deliver focused ultrasound energy below the surface of the skin.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to demonstrate the effectiveness of the Ulthera® System for non-invasive treatment to reduce wrinkles around the eyes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years.
* Subject in good health.
* Mild to moderate rhytids in the periorbital region.
* Willingness and ability to comply with protocol requirements and return for follow-up visits.
* Not pregnant.
* Provide written informed consent and HIPAA authorization.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the face.
* Deep wrinkles, numerous lines, with or without redundant skin in the area to be treated.
* Excessive hooding, with or without redundant skin, in the areas to be treated.
* Significant scarring in areas to be treated.
* Significant open facial wounds or lesions.
* Severe or cystic acne on the face.
* Presence of a metal stent or implant in the facial area to be treated.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weiss, M.D., Principal Investigator — MD Laser Skin & Vein Institute; Brian Biesman, M.D., Principal Investigator — The Nashville Centre for Laser and Facial Surgery
Locations (2):
- United States (2):
  - MD Laser Skin & Vein Institute, Hunt Valley, Maryland
  - The Nashville Centre for Laser and Facial Surgery, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-eight subjects were enrolled at two aesthetic medical facilities. Study recruitment was initiated on March 3, 2011, and concluded on July 13, 2011. Forty-five subjects were enrolled at one study site; 23 subjects were enrolled at the second study site.
Pre-assignment Details: Subjects presenting with rhytids and skin laxity in the periorbital region, Fitzpatrick Wrinkle Classification Scale (FWCS)of 3 to 7, qualified for study participation. Note: A protocol amendment restricting enrollment to FWCS scores of 3-7 occurred after 19 subjects with FWCS = 2 had been enrolled.
Groups:
- Treated Subjects: The FWCS, a 9 point scale used to classify wrinkle severity, was used to qualify subjects for study participation.
  Score 1-3 = Fine wrinkles; 4-6 = Fine to moderate-depth wrinkles, moderate number of lines; 7-9 = Fine to deep wrinkles, Numerous lines with or without redundant skin folds.
  All study subjects received an Ulthera treatment to the upper face.
Period: Overall Study
Arm/Group | Treated Subjects
Started | 68
Completed | 61
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: Adults between 30 and 65 years of age who provided informed consent and who met the inclusion/exclusion criteria and required infraorbital, lateral orbit, and brow regions to be treated bilaterally.
Groups:
- Treated Subjects: All study subjects received an Ulthera treatment to the upper face.
Arm/Group | Treated Subjects
Number analyzed (Participants) | 68
Age, Continuous [Mean (Full Range); unit: years]
  Mean (Full Range) | 51 [36 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 66
  African American/Black | 1
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 68
Fitzpatrick Skin Type [Number; unit: participants] — Skin Type I = White;very fair,red or blonde hair blue eyes;freckles;Always burns, never tans
  Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes;Usually burns, tans with difficulty
  Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans
  Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease
  Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily
  Skin Type VI = Black; Never burns, tans very easily
  participants
    Skin Type I | 0
    Skin Type II | 18
    Skin Type III | 48
    Skin Type IV | 1
    Skin Type V | 1
    Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Improvement in Periorbital Wrinkles and Rhytids Around the Eyes
Description: Improvement in periorbital skin laxity and rhytids as determined by masked assessor review of photographs at 90days post-treatment compared to baseline.
Time Frame: 90 days post-treatment
Population: Primary endpoint: Three masked assessors reviewed pre- and 90 days post-treatment photos, assessing each eye separately. 41 right, 42 left eye photos were found to be usable. Photos excluded had photographic lighting, focus and exposure inconsistencies obscuring key physical details making pre- vs. post-treatment photo comparisons impossible.
Measure: Number; unit: percentage of participants improved
Groups:
- Subjects Treated: All study subjects received an Ulthera treatment to the upper face.
Arm/Group | Subjects Treated
Number analyzed (Participants) | 64
percentage of participants improved
  Left Eye (1.5mm Transducer) | 47
  Right Eye (1.0mm Transducer) | 50

2. Secondary Outcome: Improvement in Periorbital Wrinkles and Rhytids Around the Eyes at 60 Days Post-treatment
Description: At 60 days post-treatment, each site investigator and each subject completed a Global Aesthetic Improvement Scale (GAIS), comparing with pre-treatment photos. The GAIS is 5-point scale (1-5) describing an overall assessment as follows:
  1. = Very Much Improved
  2. = Much Improved
  3. = Improved
  4. = No Change
  5. = Worse
  "Any Improvement" includes subjects assessed in categories 1-3.
Time Frame: 60 days post-treatment
Population: At 60 days, the PI and subject completed a GAIS (PGAIS and SGAIS, respectively)for comparison to pre-treatment.
Measure: Number; unit: percentage of participants improved
Groups:
- Subjects Treated: All study subject received an Ulthera treatment to the upper face.
Arm/Group | Subjects Treated
Number analyzed (Participants) | 66
percentage of participants improved
  PGAIS - Improved to Very Much Improved | 60.6
  SGAIS - Improved to Very Much Improved | 66.7

3. Secondary Outcome: Improvement in Periorbital Wrinkles and Rhytids Around the Eyes at 90 Days Post-treatment
Description: At 90 days post-treatment, each site investigator and each subject completed a Global Aesthetic Improvement Scale (GAIS), comparing with pre-treatment photos. The GAIS is 5-point scale (1-5) describing an overall assessment as follows:
  1. = Very Much Improved
  2. = Much Improved
  3. = Improved
  4. = No Change
  5. = Worse
  "Any Improvement" includes subjects assessed in categories 1-3.
Time Frame: 90 days post-treatment
Population: Data analysis was based on participants who completed a Subject Global Aesthetic Improvement scale (SGAIS) and were assessed by a study investigator via completion of a Physician Global Aesthetic Improvement scale (PGAIS)at 90 days post-treatment, per protocol.
Measure: Number; unit: percentage of participants improved
Arm/Group | Subjects Treated
Number analyzed (Participants) | 67
percentage of participants improved
  PGAIS - Improved to Very Much Improved | 59.7
  SGAIS - Improved to Very Much Improved | 67.2

4. Secondary Outcome: Improvement in Periorbital Wrinkles and Rhytids Around the Eyes at 180 Days Post-treatment
Description: At 180 days post-treatment, each site investigator and each subject completed a Global Aesthetic Improvement Scale (GAIS), comparing with pre-treatment photos. The GAIS is 5-point scale (1-5) describing an overall assessment as follows:
  1. = Very Much Improved
  2. = Much Improved
  3. = Improved
  4. = No Change
  5. = Worse
  "Any Improvement" includes subjects assessed in categories 1-3.
Time Frame: 180 days post-treatment
Population: Data analysis was based on participants who completed a Subject Global Aesthetic Improvement scale (SGAIS) and were assessed by a study investigator via completion of a Physician Global Aesthetic Improvement scale (PGAIS)at 180 days post-treatment, per protocol.
Measure: Number; unit: percentage of participants improved
Arm/Group | Subjects Treated
Number analyzed (Participants) | 61
percentage of participants improved
  PGAIS - Improved to Very Much Improved | 77.0
  SGAIS - Improved to Very Much Improved | 68.9

5. Secondary Outcome: Patient Satisfaction Questionnaire 90 Days Post-treatment
Description: Subject satisfaction determined by scores on a patient satisfaction questionnaire at 90 days post-treatment.
Time Frame: 90 days post-treatment
Population: Data analyzed included subjects completing a 90 day visit and a questionnaire assessing treatment satisfaction, comparing pre-treatment and day 90 post-treatment photographic images. Responses were tabulated.
Measure: Number; unit: percentage of participants Satisfied
Arm/Group | Subjects Treated
Number analyzed (Participants) | 67
percentage of participants Satisfied | 77.6

6. Secondary Outcome: Patient Satisfaction Questionnaire at 180 Days Post-treatment
Description: Subject satisfaction determined by scores on a patient satisfaction questionnaire at 180 days post-treatment.
Time Frame: 180 days post-treatment
Population: Data analyzed included subjects completing a 180 day visit and a questionnaire assessing treatment satisfaction, comparing pre-treatment and day 180 post-treatment photographic images. Responses were tabulated. 60 of 61 subjects provided responses. One subject's response was missing.
Measure: Number; unit: percentage of participants Satisfied
Arm/Group | Treated Subjects
Number analyzed (Participants) | 60
percentage of participants Satisfied | 72.1

7. Other Pre Specified Outcome: Subject Assessment of Pain
Description: Subjects' sensory responses to the treatment exposures were recorded for each anatomical region treated using a validated Numeric Rating Scale, 0-10, where 0 = no pain and 10 = worse pain possible.
Time Frame: Average pain scores reported during study treatment
Population: The subjects' sensory responses to the treatment exposures were recorded for each anatomical region treated, using a validated numeric rating scale of 0-10 with 1 representing no pain and 10 representing the highest degree of pain.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treated Subjects
Number analyzed (Participants) | 68
units on a scale
  Brow pain score | 5.5 [0 to 10]
  Lateral Orbit pain score | 4.8 [0 to 10]
  Infraorbit pain score | 4.3 [0 to 10]

ADVERSE EVENTS:
Arm/Group | Treated Subjects
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 5/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=68)
Visible Treatment Lines (Skin and subcutaneous tissue disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
FWCS scores assessed globally, not per eye, leading to limited data for analysis.

FWCS protocol amended to 3+ after enrollment of 19 subjects with FWCS of 2.

Unacceptable lighting, focus, exposure making some photos impossible to evaluate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No